CLINICAL TRIAL: NCT03534245
Title: Investigating Vector-borne Determinants of Aedes-transmitted Arboviral Infections in Cambodia: An Observational Longitudinal Cohort Study in Children
Brief Title: Investigating Vector-Borne Determinants of Aedes Transmitted Arboviral Infections in Cambodia: An Observational Longitudinal Cohort Study in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918100; 18-I-N100
Record Dates: First submitted 2018-05-22; First posted 2018-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08-05

CONDITIONS: Dengue Fever
Keywords: Mosquito Salivary Protein; Dengue Fever; Zika; Chikungunya; Kampong Speu; Natural History
MeSH Terms: conditions — Dengue; Zika Virus Infection; Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy children aged 2 - 9 years

SUMMARY:
Background:

Some mosquitos carry viruses that can cause disease. Some examples are dengue and Zika. The mosquitos spread disease by biting people and infecting them with the virus. Children, elderly people, and people who are already sick are especially likely to get infected. Researchers want to learn more to help make new medicines to treat these viral infections.

Objective:

To learn more about how mosquitos infect people, and why young children are more likely to get sick than other people.

Eligibility:

Healthy children 2-9 years old who live near the study site. This is Kampong Speu District Referral Hospital in Chbar Mon, Cambodia.

Design:

At visit 1, participants will have a physical exam. A small amount of blood will be taken from their arm or finger. Parents will answer questions about the participant s general health and medical history.

Participants will come back to the study site every wet season and every dry season for the next 3 years. The visits will be the same as visit 1 and take about 1 hour.

If at any time during the study the participant gets a fever and has other symptoms that could be caused by these viral diseases, they should be brought to the study site. These symptoms might include headache, pain behind the eyes, muscle pain, or joint pain. They can also include a rash that lasts longer than 12 hours.

Participation ends after the final study visit in late 2021.

DETAILED DESCRIPTION:
Mosquito-borne viruses continue to cause significant global morbidity and mortality, particularly in Southeast Asia. When mosquitoes deliver the virus into the skin of humans while probing for a blood meal, they deposit also saliva, which contains a myriad of pharmacologically active compounds that modulate the host immune system. Most vaccines against vector-borne diseases under development ignore the importance of the complex infectious inoculum delivered by the mosquito vector and the subsequent host immune response to mosquito salivary proteins. Many studies of vector-borne disease do not evaluate what role vector-derived factors play in the host immune response of these infections. A cumulative body of evidence from animal models and limited retrospective human data demonstrates that a variety of vector-derived components, including salivary components, are codelivered with the pathogen and may play an important role in the establishment and dissemination of arboviral infection. Knowledge of the effect of these vector-derived factors on the development of arboviruses in the human is limited. Here, we will establish and follow a longitudinal pediatric cohort study to describe the burden of dengue virus and to carefully examine the immune response to exposure of the salivary proteins of Aedes aegypti, the mosquito vector of dengue, Zika and chikungunya viruses. This study will serve as a foundation so that future studies may contribute to further understanding how saliva immunity impacts arboviral disease development i Cambodia, a country endemic to these viruses.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 2-9 years
4. Live within approximately 5.5 km of study site
5. In good general health as evidenced by medical history
6. Willing to allow biological samples to be stored for future research.

EXCLUSION CRITERIA:

1. Current or prior use within last 6 months of any immunosuppression (e.g. intravenous immunoglobulin, steroids, interferon therapy)
2. Treatment with another investigational drug, vaccine, or other intervention within six months of screening

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community-based cohort of children from the town of Chbar Mon in Kampong Speu, Cambodia, who live within 5.5 km to the Kampong Speu District Referral Hospital.@@@
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of symptomatic and inapparent dengue infection (serotypes 1-4) as detected semiannually via ELISA assay (binary outcome present/absent) over a three-year period in Kampong Speu in children aged 2-9 years old | Semi-Annual visits and sick/convalescent visits throughout study enrollment
  Detailed knowledge of dengue seroprevalence and transmission season variability will help establish an epidemiological foundation to prepare for larger future studies such as disease incidence studies or vector interventional trials.
Prevalence of Aedes aegypti salivary gland homogenate reactivity as detected by ELISA assay (binary outcome present/absent) during wet and dry seasons over a three-year period in Kampong Speu in children aged 2-9 years old | Semi-annual visits and sick/convalescent visits throughout study enrollment
  Characterizing the Ae. aegypti salivary protein reactivity profile in Cambodians is the first step prior to assessing how Ae. aegypti saliva exposure modulates disease in humans.

SECONDARY OUTCOMES:
Western blot analysis of sera from participants with strongest ELISA positivity to Ae. aegypti whole salivary gland homogenate compared to Anopheles and Culex to assess cross-reactive immunogenicity to mosquito saliva versus specific Aedes marke... | Semi-annual visits and sick/convalescent visits throughout study enrollment
  This next layer of analysis to identify specific immune dominant molecules, from a whole-protein approach, will provide the highestprobability of identifying novel proteins, irrespective of immune-modulatory function, that can then be characterized. It is essentialto assess reactivity to the saliva of Anopheles and Culex in order to exclude crossreactive antigens and select for Aedes-specific markers.
Positive RT-PCR result for diagnosis of dengue, chikungunya, and Zika viruses (or IgM capture ELISAs for dengue as needed) | Semi-annual visits and sick/convalescent visits throughout study enrollment
  Dengue is the predominant flavivirus, but other circulating arbovirusescomplicate the serologic diagnosis of prior immunity and it will be important to characterize this burden given the ease and little costadded to run the multiplex RT-PCR compared to a DENV RT-PCR alone. Depending upon local transmission patterns, this could informwhether additional serological assays (e.g. plaque reduction neutralization assays [PRNTs]) may be needed to assess ZIKV, CHIKV, and Culex-transmitted JEV seroprevalence. The study is not powered to detect incidence of these symptomatic Aedestransmitted disease because it would require thousands and thousands of children.
Geographic information system with all data components (mosquito catch sites, houses, schools) referenced by latitude and longitude in addition to a series of map layers (point maps, smoothed maps) to evaluate relationships between IgG intensity... | Semi-annual visits and sick/convalescent visits throughout study enrollment
  These data and analyses will allow for detailed spatiotemporal analysis of the data at individual, house and community levels. Similar published methods (except different entomological indices) were used for assessment of Anopheles salivary protein exposure at the Thai-Burma border for risk of malaria transmission.
Seroconversion to Ae. aegypti salivary homogenate in relationship to season (wet versus dry) and collected time-dependent variables defined as mean and maximum rainfall, temperature and humidity inaddition to monthly fingerpricks to evaluate ... | Semi-annual visits and sick/convalescent visits throughout study enrollment
  Assessing the persistence of anti-saliva antibody response in the dry season is critical to a biomonitoring strategy to inform future vector control programs in the area. The natural time course of salivary protein exposure, particularly in confirmed arboviral disease settings,has not been wellcharacterized. Retrospective repeat analyses of nondiseased samples have suggested that salivary IgG antibodies may last 30-40 days. 10 Seasonal variation and climate factors are implicated in both disease transmission and vector abundance.
Capture a minimum of 25 female Aedes aegypti mosquitoes for transcriptional comparison to LMVR-reared Aedes aegypti mosquitoes | Duration of study enrollment
  Wild-caught Ae. aegypti may harbor considerable difference to inbred mosquito strains maintained in insectaries. Differences in salivary and midgut composition may help explain unique vector competence aspects and immunogenicity of the strains of Ae. aegypti in Cambodia.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz F Oliveira, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Kampong Speu Referral Hospital, Chbar Mon, Kampong Speu, Cambodia

REFERENCES:
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Pingen M, Bryden SR, Pondeville E, Schnettler E, Kohl A, Merits A, Fazakerley JK, Graham GJ, McKimmie CS. Host Inflammatory Response to Mosquito Bites Enhances the Severity of Arbovirus Infection. Immunity. 2016 Jun 21;44(6):1455-69. doi: 10.1016/j.immuni.2016.06.002. PMID 27332734
- [Background] Machain-Williams C, Mammen MP Jr, Zeidner NS, Beaty BJ, Prenni JE, Nisalak A, Blair CD. Association of human immune response to Aedes aegypti salivary proteins with dengue disease severity. Parasite Immunol. 2012 Jan;34(1):15-22. doi: 10.1111/j.1365-3024.2011.01339.x. PMID 21995849
- [Derived] Odio CD, Yek C, Hasund CM, Man S, Ly P, Nhek S, Chea S, Lon C, Voirin C, Huy R, Leang R, Huch C, Lamirande EW, Whitehead SS, Oliveira F, Manning JE, Katzelnick LC. Immunity to Non-Dengue Flaviviruses Impacts Dengue Virus Immunoglobulin G Enzyme-Linked Immunosorbent Assay Specificity in Cambodia. J Infect Dis. 2025 Feb 20;231(2):e337-e344. doi: 10.1093/infdis/jiae422. PMID 39297691
- [Derived] Manning JE, Chea S, Parker DM, Bohl JA, Lay S, Mateja A, Man S, Nhek S, Ponce A, Sreng S, Kong D, Kimsan S, Meneses C, Fay MP, Suon S, Huy R, Lon C, Leang R, Oliveira F. Development of Inapparent Dengue Associated With Increased Antibody Levels to Aedes aegypti Salivary Proteins: A Longitudinal Dengue Cohort in Cambodia. J Infect Dis. 2022 Oct 17;226(8):1327-1337. doi: 10.1093/infdis/jiab541. PMID 34718636
- [Derived] Manning JE, Oliveira F, Parker DM, Amaratunga C, Kong D, Man S, Sreng S, Lay S, Nang K, Kimsan S, Sokha L, Kamhawi S, Fay MP, Suon S, Ruhl P, Ackerman H, Huy R, Wellems TE, Valenzuela JG, Leang R. The PAGODAS protocol: pediatric assessment group of dengue and Aedes saliva protocol to investigate vector-borne determinants of Aedes-transmitted arboviral infections in Cambodia. Parasit Vectors. 2018 Dec 20;11(1):664. doi: 10.1186/s13071-018-3224-7. PMID 30572920